CLINICAL TRIAL: NCT01690481
Title: Neurocognitive and Neuroanatomical Studies in Young Children With Type 1 Diabetes Mellitus
Brief Title: The Effects of High and Low Blood Glucose Values on the Brain in Children With Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: William E And Aenid R Weisgerber Foundation (Other)
Responsible Party: Principal Investigator, Tandy Aye, Assistant Professor, Stanford University
Other Study IDs: SU-09242009-4020; IRB# 7723
Record Dates: First submitted 2012-08-06; First posted 2012-09-21 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Simplified Brochure

Neuropsychological Testing/Assessment is like games for the child. They are asked to complete the sequence, identify pictures, explain what is happening, etc. There is no personality testing involved. Part of the standard IQ testing is done but no IQ score is obtained. Age appropriate testing is done for each child.

The MRI is an enclosed machine. We have the child sit in a simulator after the neuropsychological testing to see what it will be like, including the sounds, etc. You will be given a video about MRI testing to view as well. The staff that does this has been doing this for years in a wide variety of children, young, developmental delayed, etc. The staff does this WITHOUT sedation. Some children cannot sit still through the entire series. We need to get six, 10 minute scans. Children are allowed movement such as the need to wiggle their toes and move in between each scan.

The Neuropsychological Testing can be scheduled in the late afternoons if it is more convenient for your family. This visit may take 3-4 hours. The MRI scanning can be scheduled after 5pm and may take up to 2 hours depending on the child's cooperation. You maybe asked to repeat the Neuropsychological Testing and MRI scanning 24 months later.

DETAILED DESCRIPTION:
BROCHURE:

Name of Study: Neuropsychological and Neuroanatomical Studies in Young Children Study Directors: Tandy Aye, MD; Bruce Buckingham, MD; Darrell Wilson, MD

About the Study: This study is being conducted to see if Type 1 diabetes mellitus has any affect on learning, behavior and development in young children. Fifty to 60 children between the ages of 3 to less than 10 years with Type 1 diabetes mellitus will have neuropsychological testing and a nonsedated MRI scan of the head performed. The study will compare the results from those with diabetes to a control group of 20-30 children between the ages of 3 to less than 10 years without Type 1 diabetes mellitus. The control subjects will have neuropsychological testing and a nonsedated MRI scan of the head performed as well. All subjects maybe asked to repeat the neuropsychological testing and nonsedated MRI scan of the head 24 months later. The children with Type 1 diabetes mellitus will not have any changes made to their current diabetes regimen. The children with Type 1 diabetes mellitus should continue to check blood glucose values as required by their doctors and bring their meter(s) for downloading to each visit. The child should also tell his/her doctor about the frequency of severe low and high blood glucose values to his/er doctor as routinely asked.

Participant Schedule:

1. One visit for 3-4 hours at the Stanford Medical Center to complete neuropsychological testing and to become familiar with the MRI scanner.
2. Subjects who need to become more familiar with the MRI scanning process will view a video tape at home.
3. One visit for 1-2 hours at Stanford Medical Center to have the MRI scan of the head completed.
4. Subjects may have the neuropsychological testing and MRI scan repeated 24 months from time of the initial testing and scan.

Inclusion Criteria:

To take part in the study, the child must meet the following inclusion criteria:

1. Be between the ages of 3 to 10 years.
2. Have been diagnosed with type 1 diabetes for at least 6 months.
3. Do not have plans to move out of the area within the next 36 months.

Exclusion Criteria:

A history of head trauma with any loss of consciousness cystic fibrosis prematurity (born less than 30 weeks of gestation) significant developmental delay (lack of single word speech or ability to walk independently by 18 months of age) neurologic disease independent of diabetes (eg seizure disorder or medical contraindication to MRI procedure (eg metal appliances such as braces).

Compensation: There will be no cost to the subjects to participate in this research study. Participants will be compensated for their time. If you are interested in participating in this study and you meet the inclusion criteria, please contact:

Kim Caswell, APRN, BC (650)-724-1201 Email: kcaswell@stanford.edu Tandy Aye, MD (650)-723-5791 Email: taye@stanford.edu

ELIGIBILITY:
Inclusion Criteria:

* To take part in the study, you or your child must meet the following inclusion criteria:

  * Be between the ages of 3 to 10 years.
  * Have been diagnosed with type 1 diabetes for at least 6 months.
  * Do not have plans to move out of the area within the next 36 months.

Exclusion Criteria:

If the interested participant has a history of:

* head trauma with any loss of consciousness,
* cystic fibrosis,
* prematurity (born less than 30 weeks of gestation),
* significant developmental delay (lack of single word speech or ability to walk independently by 18 months of age),
* neurologic disease independent of diabetes (eg seizure disorder or medical contraindication to MRI procedure (eg metal appliances such as braces)

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children between ages 3 to 10 with and without type 1 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2006-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
MRI brain volumes | 3 years

SECONDARY OUTCOMES:
Neuropsychological scores | 3 yr
  FSIQ, Memory score, Verbal comprehension score

CONTACTS AND LOCATIONS:
Overall Officials: Tandy Aye MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States